CLINICAL TRIAL: NCT05440877
Title: Efficacy of Virtual Reality (VR) Video-based Learning for Enhancing Nursing Students' Self-efficacy in Delivering Smoking Cessation Intervention: A Randomized Controlled Trial
Brief Title: Virtual Reality Video-based Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VR_smoking
Record Dates: First submitted 2020-03-01; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Smoking Cessation; Nursing Education
Keywords: Virtual reality; Nursing; Smoking
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Individual randomization by serially numbered opaque sealed envelope (SNOSE) will be used to ensure the allocation sequence was concealed from both course teacher and participants before the group allocation. he participants will know the trial group and discussion group allocation by opening an envelop after they submit the consent form. All pre-post questionnaires are anonymous. All participants will be concealed of group allocation before consent, but they will not be blinded of the intervention. Two specialists in smoking cessation who will mark the group assignment will be blinded to group allocation of all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Provided with a tutorial guide, and VR-based teaching materials in the tutorial session
  Interventions: Behavioral: VR materials; Behavioral: Tutorial guide
- Control group (Experimental): Provided with the tutorial guide in the tutorial session.
  Interventions: Behavioral: Tutorial guide

INTERVENTIONS:
Behavioral: VR materials — In the lecture room for the intervention group, participants in the intervention group will be given QR codes for viewing these online videos and VR cardboards, a web including photo hunt sections that allow viewers to find cues for smoking cessation treatment. They are asked to view these videos and photos with their own mobile phones.
  Arms: Intervention group
Behavioral: Tutorial guide — A tutorial guide including description of the smokers' cases

SUMMARY:
This teaching development aims to enhance the clinical reasoning and empathy of nursing students in nursing students in smoking cessation training. The evaluation aims to assess the feasibility and efficacy of virtual reality (VR) video-based learning for enhancing self-efficacy in delivering smoking cessation intervention. The proposed study is 2-arm, waitlist-control, pragmatic randomized controlled trial (RCT) (allocation ratio 1:1), by comparing the self-efficacy and performance of clinical reasoning between nursing students who are provided VR videos of a smoker's real-life scenario and reading materials (intervention group) and those who are only provided the same reading materials (control). Individual randomization will be used. All participants will be given a group assignment and expected to complete the assignment by the end of the tutorial. The group assignment and self-administered pre- and post-learning survey will be used for the teaching outcome evaluation.

DETAILED DESCRIPTION:
The proposed study is 2-arm, waitlist-control, pragmatic randomized controlled trial (RCT) (allocation ratio 1:1), by comparing the self-efficacy and performance of clinical reasoning between nursing students who are provided VR videos of a smoker's real-life scenario and reading materials (intervention group) and those who are only provided the same reading materials (control). Individual randomization will be used. All participants will be given a group assignment and expected to complete the assignment by the end of the tutorial. The group assignment and self-administered pre- and post-learning survey will be used for the teaching outcome evaluation.

ELIGIBILITY:
Inclusion Criteria:

The study targets to recruit candidates of Master of Nursing who are taking the course "Tobacco Dependency Nursing Intervention and Management (NURS8205)" (n=65). All candidates are registered nurses.

Exclusion Criteria:

Students who cannot understand Cantonese will be excluded from the trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Self-efficacy in delivering smoking cessation intervention | Before and after the tutorial (at 1-day)
  (1) Understand the quitting barriers of smokers barriers; (2) Design quit plan for smoking patients; (3) Prioritize interventions for smoking patients; (4) Educate smoking patients on essential tasks; (5) Overall confidence in the management of smoking patients; and (6) Overall competence in the management of smoking patients. Each item can be scored from 0 (not at all competent) to 10 (extremely competent).
Empathy in delivering smoking cessation intervention | Before and after the tutorial (at 1-day)
  (1) Show empathy to smoking patients; (2) Show care to smoking patients; (3) Being positive; (4) See things from smokers' perspective; (5) Can you show tender feeling for smokers? (0: Not at all, 5: half and half, 10: extremely); (6) Do you feel sorry for smokers who are unable to quit? (0: Not sorry at all, 5: half and half, 10: extremely sorry); (7) Do you feel sorry for smokers who do not want to quit? (0: Not sorry at all, 5: half and half, 10: extremely sorry); and (8) Do you feel annoyed if smokers ignore your cessation advice (0: Not annoyed at all, 5: half and half, 10: extremely annoyed). Each item can be scored from 0 (not at all competent) to 10 (extremely competent).
Lasater Clinical Judgment Rubric | After the tutorial (at 1-day)
  (1) Effective noticing: Focused observation; (2) Effective noticing: Recognizing deviations from expected patterns; (3) Effective noticing: Information seeking; (4) Effective interpreting: Prioritizing data; (5) Effective interpreting: Making sense of data; (6) Effective responding: Well-planned intervention/flexibility; (7) Effective responding: Being skilful; (8) Effective reflecting: Evaluation/self-analysis. Each item can be scored from exemplary, accomplished, developing and beginning.

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Derek Y Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The study information can be provided upon requests made to the principle investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 5 years
Access Criteria: For non-commercial purpose.

REFERENCES:
- [Derived] Cheung YTD, Zhang G, Luk TT, Zhang M, Lam VSF, Chan MMK, Wang MP, Chan SSC. Effect of narrative videos and mini-VR games in nursing smoking cessation training on empathy and self-efficacy of smoking cessation counseling: A randomized controlled trial. Nurse Educ Today. 2024 Sep;140:106272. doi: 10.1016/j.nedt.2024.106272. Epub 2024 Jun 4. PMID 38851019